CLINICAL TRIAL: NCT05636930
Title: To Evaluate the Accuracy of Sleep Parameters Evaluated by Wearable Sleep Devices
Brief Title: Accuracy Assessment of Sleep Monitoring Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanshan Lu (Other)
Responsible Party: Sponsor-Investigator, Shanshan Lu, Doctor of Medicine(M.D.), Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2002(052)
Record Dates: First submitted 2022-10-26; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Wearable Devices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- smart bracelet: Type and specification:FRA-B39
  Interventions: Other: Test the accuracy of the wearable device

INTERVENTIONS:
Other: Test the accuracy of the wearable device — No intervention was done for the subjects

SUMMARY:
As a necessary process of life, sleep is an important link for the body to recover, integrate and consolidate memory. However, the fast pace of life in modern society and people's bad living habits are easy to cause sleep disorders. Sleep disorders are often the main factors that induce or aggravate cardiovascular and cerebrovascular diseases. Sleep staging is an important basis for sleep quality assessment and related disease diagnosis. At present, electroencephalography (EEG) has become the gold standard for judging sleep stages. However, this kind of method requires long-term contact of multiple electrodes with the human body, which is easy to affect the natural sleep of the subjects, so it is not suitable for sleep monitoring in home environment. Studies have shown that sleep is related to the regulation of autonomic nervous system, and heart rate variability (HRV) in sleep also shows periodic changes similar to brain waves. Smartwatch/bracelet can continuously monitor the user's pulse wave and acceleration data comfortably and without feeling. HRV features can be extracted using pulse wave data, and then sleep staging can be realized based on the correlation between HRV and brain waves, and sleep quality can be evaluated. Therefore, healthy sleep research aims to use smart devices to achieve sleep monitoring in the home environment and improve people's sleep quality

ELIGIBILITY:
Inclusion Criteria:

* a. Adults aged 18 and above and under the age of 60; The age of the subjects was divided into two age groups: 18-44, 45-60, and the ratio between the two groups was 1:1.2-1:0.8. The ratio of female to male is between 1:1.1 and 1:1.0; b. No patients with serious cardiovascular and cerebrovascular diseases, moderate degree of depression, anxiety disorder or severe apnea; HAMD<=20;HAMA <=13;AHI< 30 c. Subjects did not drink alcohol or take sleep intervention drugs during the program; d. People with sleep disorders and insomnia can be included in the subjects, but the total number is no more than 50%, and should be clearly marked; e. Having Chinese nationality and residing in China; f. Agree to be monitored by PSG and wear wearable devices; Voluntary entry, informed consent or consent to privacy agreement.

Exclusion Criteria:

* a. Patients with a history of depression, anxiety and other mental disorders; HAMD>20;HAMA>13 b. Patients with existing atherosclerotic cardiovascular diseases, such as coronary heart disease and severe peripheral atherosclerotic disease; c. age >60 d. Patients with obstructive sleep apnea (AHI >30); Use of drugs or substances affecting the central nervous system in the preceding 2 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: china
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of sleep parameters of wearable devices | 8-10AM
  Sleep Latency,sleep efficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Shanshan Lu, Jinan, Shandong, China